CLINICAL TRIAL: NCT04082871
Title: Assessing the Impact of Medication Management Review Service for Females Diagnosed With Depression and Anxiety
Brief Title: Medication Review in Women With Depression and Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Applied Science Private University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1IRB/2016/04
Record Dates: First submitted 2019-09-02; First posted 2019-09-09 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: Depression, Anxiety; Adherence, Patient
Keywords: Medication management review service; Pharmaceutical care; Clinical pharmacist
MeSH Terms: conditions — Depression; Anxiety Disorders; Patient Compliance

STUDY DESIGN:
Intervention Model Description: Following recruitment, participants were randomized into two groups (1:1 randomization), active and control, using the computer-generated randomization program (www.randomization.com). The researcher generated the allocation sequence, and assigned the participants to their group. Participant who came into the clinic during the clinic's working hours (Sunday to Thursday, from 9 am to 1 pm) were approached consecutively and allocated to the active or control group. Participants were not aware of which study group they were assigned to; only the researcher was aware of each patient's group assignment.
  Participants in the active and control groups completed a baseline and follow-up (3 months from baseline) visits at the same outpatient psychiatric clinic with the researcher conducting the interview using the study tool to complete the MMR process.
Who Masked: Participant
Masking Description: This single-blind parallel randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): All pharmacist level counseling and education regarding treatment, adherence and self-care activities were delivered to the active group patients only (planned to take 15 minutes). Patient level TRPs (any TRP that could be resolved via patient education and counseling) were resolved directly with the patient by the clinical pharmacist.
  A letter with the identified TRPs (prioritized from most important to least important) for each patient in the active group was sent to the patient's psychiatrist by the researcher in sealed envelopes. The psychiatrist either accepted or rejected the recommendations. In case the recommendations were accepted, the psychiatrist implemented the recommended changes. Patients were informed by a phone call by the pharmacist to visit their psychiatrist soon after the recommendations were approved for the changes to be applied.
  If the recommendations were rejected, the psychiatrist stated the reason of rejection and discussed it with the pharmacist.
  Interventions: Other: Medication management review
- Control (Active Comparator): Control group patients also underwent the baseline interview with the researcher at the psychiatric clinic, TRPs were identified and documented. No intervention was provided by the pharmacist and no letter was sent to the patients' psychiatrists. In case a patient was found to have a life-threatening TRP, the patient was excluded from the study and reported to the psychiatrist due to ethical considerations.
  After study completion, all patients in the control group received the MMR service, and a letter with their TRPs and recommendations to resolve them was sent by the pharmacist to their psychologist
  Interventions: Other: Medication management review

INTERVENTIONS:
Other: Medication management review — The researcher screened each completed an MMR template and verified that all information in each patient template was complete. A classification system was then used to identify the TRPs which either actually or potentially interfered with the clinical outcomes for each patient.[19] This system was explained in detail and applied successfully in many previous studies.[10, 14, 20] The researcher then identified TRPs for each patient in both groups using evidence-based medicine. The TRPs including unneeded drug treatment, untreated condition/s, efficacy/effectiveness issues, safety issues, inadequate knowledge, inappropriate adherence to pharmacological therapy, inappropriate adherence to self-care activities and miscellaneous problems.

SUMMARY:
This study sought to assess the impact of the MMR service on identifying and resolving TRPs, improving adherence, depression and anxiety scores in females diagnosed with depression and anxiety in Jordan

DETAILED DESCRIPTION:
Participants were recruited into this single-blind parallel randomized controlled trial and randomized into active and control groups. A clinical pharmacist identified TRPs for all participants. Adherence, depression and anxiety scores were assessed. Active group patients received the MMR service: pharmacist-delivered counseling and a letter with recommended changes in the patient's treatment plan was sent to the patient's psychiatrist to be applied. Control group participants did not receive the intervention. Follow-up assessments were completed for all patients at 3 months from baseline. Main outcome measures were TRPs, adherence, depression and anxiety scores.

ELIGIBILITY:
Inclusion Criteria:

* Jordanian females or residents in Jordan for the last 12 months and planning to stay in Jordan for 6 months (the study follow-up period),
* above the age of 18 years
* diagnosed with depression and/or anxiety for at least 4 weeks duration
* taking medications for depression and/or anxiety

Exclusion Criteria:

* presence of a cognitive problem or sensory impairment which may prevent communication with the patient (reported by the patient's psychiatrist)
* being not able to speak or write Arabic (reported by the patient)

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Females diagnosed with depression and/or anxiety and attending the psychiatric clinics at Jordan University Hospital (JUH)
Enrollment: 73 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-01-10 (Actual)

PRIMARY OUTCOMES:
Evaluate the effect of the medication management review service delivered to females living in Jordan and diagnosed with depression and anxiety | 6 months
  the medication management review service will be measured by the reduction of treatment related number after providing the service

SECONDARY OUTCOMES:
Patient's satisfaction with the medication management review service | 6 months
  satisfaction will be measured by the willingness of patients to pay for the provided services

IPD SHARING:
Plan to Share IPD: Undecided